CLINICAL TRIAL: NCT02252627
Title: An Observational Study to Test the Effect of the Vasoactive Drugs Phenylephrine and Ephedrine on the Stroke Volume and Microvascular Blood Flow of Healthy Volunteers
Brief Title: The Effect of Phenylephrine and Ephedrine on Microvascular Blood Flow
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: H10102013
Record Dates: First submitted 2014-09-25; First posted 2014-09-30 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Healthy volunteers
  Interventions: Drug: Administration of phenylephrine; Other: Measurement of stroke volume; Other: Contrast enhanced ultrasound scan; Drug: Administration of ephedrine

INTERVENTIONS:
Drug: Administration of phenylephrine — Intravenous phenylephrine will be administered in 50-100 microgram increments until the mean arterial blood pressure has increased by 25% compared to baseline, or until a maximum dose of 1mg has been administered.
Other: Measurement of stroke volume — The measurement of stroke volume will be performed using an Oesophageal Doppler Monitor
Other: Contrast enhanced ultrasound scan — Microvascular blood flow will be measured using a contrast enhanced ultrasound scan
Drug: Administration of ephedrine — Intravenous ephedrine will be administered in 3-6mg increments until the mean arterial blood pressure has increased by 25% compared to baseline, or until a maximum dose of 30mg has been administered.

SUMMARY:
During operations to treat abdominal problems the blood pressure can fall, resulting in falls in blood flow to the vital organs. This fall can be treated by the administration of drugs that cause constriction of blood vessels. Although these drugs correct falls in blood pressure, it is unclear what effect they have on blood flow from the heart and to the vital organs.

In this study of healthy volunteers we aim to better understand the changes in blood flow in both small and large vessels that occur in response to administration of these drugs. To do this we will use two different techniques of ultrasound imaging. A narrow (4-5mm) ultrasound probe will be inserted into the oesophagus via a nostril to measure blood flow in a major blood vessel. A second probe will rest on the abdomen and will record changes in blood flow in small vessels of the liver. Two drugs which raise the blood pressure via different mechanisms will be administered and the changes in flow from the heart and to vital organs will be measured and compared.

DETAILED DESCRIPTION:
Optimising the cardiac output is essential to ensure adequate organ perfusion in patients who are undergoing major surgery. To enable this cardiac output (CO) is frequently monitored during operations using a variety of techniques; one such technique is trans-oesophageal Doppler ultrasound also known as oesophageal Doppler monitoring (ODM). ODM measurement of CO is a less invasive technique than many currently used methods, and has recently been recommended by NICE for adoption in clinical practice. The matching of microvascular blood flow and CO is advantageous for visceral organs, in marrying demands for oxygen and nutrients to their delivery. Major surgery and the attendant requirement for general anaesthesia can result in dramatic changes in blood pressure (BP) and CO. These changes can be corrected by the administration of vasoactive drugs such as phenylephrine and ephedrine, although it is unclear what effects these drugs have on microvascular blood flow (MVBF) to the intra-abdominal viscera. Whilst they correct falls in BP, and hence may increase visceral flow, this increased BP is partially mediated via splanchnic vasoconstriction, which may result in decreased blood flow. A greater appreciation of the effect of these vasoactive drugs on the CO and MVBF may help with the development of more refined algorithms for their use in the clinical setting. In our clinical physiology laboratories we regularly employ contrast-enhanced ultrasound (CEUS) using a Phillips iU22, to measure MVBF in healthy males following a variety of physiological challenges. This minimally invasive ultrasound based imaging technique is ideal for gaining an insight into the effect various physiological interventions have on tissue blood flow and could be readily used to chart changes in visceral MVBF and CO following vasoactive drug administration. Transference of this investigative approach to a clinical setting has the potential to greatly improve the care of the surgical patient under anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years
* Male
* Able to consent in English by themselves
* Absence of any exclusion criteria

Exclusion Criteria:

* A BMI < 20 or > 28 kg•m2
* Active cardiovascular disease: uncontrolled hypertension (BP > 140/90), angina, heart failure (class III/IV), arthymia, right to left cardiac shunt or recent cardiac event
* Individuals taking alpha or beta-adrenergic blocking agents, monoamine oxidase inhibitors, tricyclic antidepressants, serotonin or noradrenaline selective reuptake inhibitors, quinidine, cardiac glycosides or buspirone (or who have ceased taking them in the previous 14 days¬)
* Cerebrovascular disease: previous stroke, aneurysm (large vessel or intracranial)
* Peripheral vascular disease
* Metabolic disease: hyper and hypo parathyroidism, untreated hyper and hypothyroidism, Cushing's disease, types 1 or 2 diabetes
* Active inflammatory bowel disease, or renal disease
* Known prostatic hypertrophy
* Malignancy
* Clotting dysfunction
* Previous oesophageal surgery
* Individuals with a known history of oesophageal varices
* Individuals with a known history of epistaxis
* Family history of early (<55y) death from cardiovascular disease
* Known sensitivity to SonoVue, ephedrine or phenylephrine
* Participants who have taken part in any other research study in the last three months which involved: taking a drug; being paid a disturbance allowance; having an invasive procedure (eg blood sample >50ml, muscle biopsies) or exposure to ionising radiation.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male volunteers
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Change in microvascular blood flow | 30 minutes
  Microvascular visceral blood flow is assessed using contrast enhanced ultrasound, and will be assessed before and after the administration of each drug.

SECONDARY OUTCOMES:
Change in stroke volume | 30 mins
  The change in stroke volume will be assessed using an Oesophageal Doppler Monitor, and will be assessed before and after the administration of each drug.

CONTACTS AND LOCATIONS:
Overall Officials: John P Williams, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, School of Medicine, Division of Medical Sciences and Graduate Entry Medicine, Derby, Derbyshire, United Kingdom